CLINICAL TRIAL: NCT01192516
Title: Effectiveness of Tailored Activity Pacing for Symptomatic Osteoarthritis
Acronym: AIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E7557-R
Record Dates: First submitted 2010-08-25; First posted 2010-09-01 (Estimated); Results first posted 2015-03-19 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-03

CONDITIONS: Osteoarthritis; Pain
Keywords: Osteoarthritis; Activity Pacing
MeSH Terms: conditions — Osteoarthritis; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental): Tailored activity pacing
  Interventions: Behavioral: Tailored Activity Pacing
- Arm 2 (Experimental): General activity pacing and symptom management (Occupational therapy)
  Interventions: Behavioral: General Activity Pacing
- Arm 3 (No Intervention): Usual care group

INTERVENTIONS:
Behavioral: Tailored Activity Pacing — Therapeutic intervention will be based on a tailored approach using collected data on symptom and activity patterns of each participant.
  Arms: Arm 1
Behavioral: General Activity Pacing — Therapeutic intervention using generalized pacing instruction to manage symptoms
  Arms: Arm 2

SUMMARY:
The primary objective of this project is to examine effectiveness of a tailored pacing intervention on fatigue, pain, and physical function compared to general pacing intervention and usual care groups. A secondary objective is to evaluate the natural history of symptoms and physical disability over time among people with knee and hip osteoarthritis.

DETAILED DESCRIPTION:
In the United States, osteoarthritis is a growing public health issue and a leading cause of disability among older adults. Almost 50% of users of the Veterans Affairs (VA) system present with osteoarthritis. Veterans are a particularly important group to target for symptom management interventions as they are twice as likely as non-veterans to report chronic joint symptoms and activity limitations. There are few evidence-based symptom management interventions offered by health care professionals, such as occupational and physical therapists, at the time when people are seeking treatment for their symptoms. The proposed activity pacing intervention is individually-tailored to a person's symptom and activity patterns. This tailoring provides a personally-relevant and focused intervention that may help people adopt this strategy into their daily lives.

ELIGIBILITY:
Inclusion Criteria:

* Age of 50 years and older
* Reported pain for at least 3 months
* Mild-moderate pain severity according to the WOMAC pain scale
* Radiographic evidence of knee or hip osteoarthritis (Kellgren-Lawrence score of 2 in at least one joint)
* Community-dwelling (i.e. own home, apartment, senior residence)
* Ambulatory with or without a cane or walker
* Adequate cognition to complete study activities (score of 5 on the 6-Item Screener)
* Ability to use the Actiwatch-S (Phillips-Respironics, Mini-Mitter, Bend OR)accelerometer to record symptoms and activity patterns (ascertained by completion of a learning module specific to the use of the device in this study)
* English-speaking

Exclusion Criteria:

* Self-reported medical history of conditions with pain and/or fatigue as a known and marked symptom (e.g multiple sclerosis, rheumatoid arthritis)
* Medically unstable (e.g. acute conditions or acute presentations of chronic conditions)
* Anemia (hemoglobin of <10 for men and <11 for women)
* Unmanaged thyroid dysfunction (Thyroid stimulating hormone <.035>5.5 mg/dl)
* 2 or more days of complete bed rest within the last month
* Limb hemiplegia or amputation
* Arthroscopic procedure within the previous 2 months
* Joint injection within the previous 3 months
* Total or partial joint replacement within the previous 6 months
* Self-reported illness or conditions that impair cooperation with the study team or ability to complete study procedures
* Current enrollee in physical or occupational therapy for symptoms associated with osteoarthritis
* Current attendance or attendance within the previous year in a cognitive behavioral therapy program or other self-management program that includes activity pacing instruction
* Any other unforeseen exclusion criteria that, by the opinion of the study personnel, would make the participant unable to safely or effectively complete the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2010-01; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan L Murphy, ScD OTR, Principal Investigator — VA Ann Arbor Healthcare System
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Murphy SL, Schepens Niemiec S, Lyden AK, Kratz AL. Pain, Fatigue, and Physical Activity in Osteoarthritis: The Moderating Effects of Pain- and Fatigue-Related Activity Interference. Arch Phys Med Rehabil. 2016 Sep;97(9 Suppl):S201-9. doi: 10.1016/j.apmr.2015.05.025. Epub 2016 May 17. PMID 27207435
- [Derived] Murphy SL, Lyden AK, Clary M, Geisser ME, Yung RL, Clauw DJ, Williams DA. Activity pacing for osteoarthritis symptom management: study design and methodology of a randomized trial testing a tailored clinical approach using accelerometers for veterans and non-veterans. BMC Musculoskelet Disord. 2011 Aug 2;12:177. doi: 10.1186/1471-2474-12-177. PMID 21810253

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential participants were recruited through fliers and advertisements.
Groups:
- Tailored Activity Pacing: Tailored Activity Pacing: Therapeutic intervention was based on a tailored approach using collected data on symptom and activity patterns of each participant.
- Usual Care Group: Participants receiving usual care
Period: Overall Study
Arm/Group | Tailored Activity Pacing | General Activity Pacing | Usual Care Group
Started | 66 (Indicates number of people initially randomized to group) | 66 (Indicates number of people initially randomized to group) | 63 (Indicates number of people initially randomized to group)
Completed | 46 | 49 | 55
Not Completed | 20 | 17 | 8
Not completed — Lost to Follow-up | 7 | 10 | 7
Not completed — Withdrawal by Subject | 4 | 4 | 1
Not completed — started new treatment | 5 | 1 | 0
Not completed — Unable to follow Actiwatch instructions | 4 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Tailored activity pacing
  Tailored Activity Pacing: Therapeutic intervention was based on a tailored approach using collected data on symptom and activity patterns of each participant.
- Arm 2: General activity pacing and symptom management
  General Activity Pacing: Therapeutic intervention using generalized pacing instruction to manage symptoms
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Total
Number analyzed (Participants) | 66 | 66 | 63 | 195
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 39 | 36 | 36 | 111
  >=65 years | 27 | 30 | 27 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (8.1) | 64.1 (8.3) | 65.8 (8.7) | 64.8 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 41 | 39 | 120
  Male | 26 | 25 | 24 | 75
Region of Enrollment [Number; unit: participants] — All participants were recruited in the Southeastern Michigan Area
  participants
    United States | 66 | 66 | 63 | 195

OUTCOME MEASURES:

1. Primary Outcome: Fatigue- Brief Fatigue Inventory (BFI)
Description: This is a summary measure of fatigue severity and fatigue interference items in which the average of 9 items is taken. Each item is rated on a scale of 0 - 10. A higher score is worse fatigue.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tailored Activity Pacing | General Activity Pacing | Usual Care Group
Number analyzed (Participants) | 66 | 66 | 63
units on a scale | 3.06 (2.34) | 3.18 (2.45) | 2.70 (2.31)

2. Primary Outcome: Fatigue-BFI
Description: This is a summary measure of fatigue severity and interference items in which the average of 9 items is taken. Each item is rated on a scale of 0 - 10. A higher score is worse fatigue.
Time Frame: 10 weeks post-baseline
Population: Sample numbers may differ due to missing data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tailored Activity Pacing | General Activity Pacing | Usual Care Group
Number analyzed (Participants) | 49 | 50 | 60
units on a scale | 3.35 (2.13) | 3.09 (2.14) | 2.98 (2.28)

3. Primary Outcome: Fatigue-BFI
Description: This is a summary measure of fatigue severity and interference items in which the average of 9 items is taken. Each item is rated on a scale of 0 - 10. A higher score indicates worse fatigue.
Time Frame: 6 months post-baseline
Population: Sample numbers may vary due to missing data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tailored Activity Pacing | General Activity Pacing | Usual Care Group
Number analyzed (Participants) | 46 | 48 | 54
units on a scale | 3.30 (2.36) | 2.90 (1.98) | 2.83 (2.26)
Statistical Analysis 1: Comparison: Tailored Activity Pacing vs General Activity Pacing vs Usual Care Group; Test type: Superiority or Other; p = .85, Mixed Models Analysis; Adjusted for age, gender, pain level, and body mass index at baseline

4. Primary Outcome: Pain- Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)
Description: This is a summary of reported pain in specific activities. It is 5 questions with answers ranging from 0 - 4. Total possible score is 20 in which a higher score is worse pain.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 63 | 66 | 63
units on a scale | 8.23 (2.99) | 8.19 (3.37) | 8.27 (3.32)

5. Primary Outcome: Pain- WOMAC
Description: This is a 5-item pain scale in which scores from 0 - 4 are summed. A higher score indicates more pain.
Time Frame: 10 weeks post-baseline
Population: Sample numbers may differ due to missing data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tailored Activity Pacing | General Activity Pacing | Usual Care Group
Number analyzed (Participants) | 49 | 50 | 60
units on a scale | 8.10 (3.43) | 7.16 (3.11) | 7.83 (3.46)

6. Primary Outcome: Pain- WOMAC
Description: This is a 5 item pain scale in which items on a scale of 0 - 4 are summed. A higher score means more pain.
Time Frame: 6 months post baseline
Population: Numbers may vary due to missing data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tailored Activity Pacing | General Activity Pacing | Usual Care Group
Number analyzed (Participants) | 47 | 49 | 54
units on a scale | 7.63 (3.57) | 7.33 (2.76) | 6.68 (3.29)
Statistical Analysis 1: Comparison: Tailored Activity Pacing vs General Activity Pacing vs Usual Care Group; Test type: Superiority or Other; p = .06, Mixed Models Analysis; Adjusted for age, gender, and body mass index

7. Secondary Outcome: Physical Function- Six Minute Walk
Description: Six minute walk is the distance (in feet) that people walk at a usual pace over 6 minutes
Time Frame: Baseline
Population: Numbers may vary due to missing data
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | Tailored Activity Pacing | General Activity Pacing | Usual Care Group
Number analyzed (Participants) | 66 | 66 | 62
feet | 1185.3 (263.3) | 1208.6 (255.2) | 1209.4 (260.1)

8. Secondary Outcome: Physical Function- Six Minute Walk
Description: This is the distance in feet that people walk over 6 minutes.
Time Frame: 10 weeks post-baseline
Population: Numbers may differ due to missing data
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | Tailored Activity Pacing | General Activity Pacing | Usual Care Group
Number analyzed (Participants) | 50 | 50 | 60
feet | 1200.5 (260.1) | 1249.4 (217.3) | 1236.1 (246.1)

9. Secondary Outcome: Physical Function- Six Minute Walk
Description: This is the distance people walk in feet over 6 minutes
Time Frame: 6 months post baseline
Population: Numbers may differ due to missing data
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | Tailored Activity Pacing | General Activity Pacing | Usual Care Group
Number analyzed (Participants) | 46 | 46 | 49
feet | 1225.4 (240.1) | 1264.3 (192.9) | 1222.4 (265.6)
Statistical Analysis 1: Comparison: Tailored Activity Pacing vs General Activity Pacing vs Usual Care Group; Test type: Superiority or Other; p = .36, Mixed Models Analysis — Adjusted for age, gender, body mass index, and pain at baseline

ADVERSE EVENTS:
Time Frame: Data were collected from baseline through completion of Time 3 outcome measures at 6 months
Arm/Group | Arm 1 | Arm 2 | Arm 3
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/66 | 0/63
Other Adverse Events (participants affected / at risk) | 3/66 | 3/66 | 1/63
OTHER ADVERSE EVENTS (reported when occurring in more than 4.55% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=66) | Arm 2 (N=66) | Arm 3 (N=63)
x-ray mistakes (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 1 (1) — most other reportable events occurred because of x-ray errors. One subject had their hips x-rayed instead of knees. Other subjects had incomplete views of their knees on xray

LIMITATIONS AND CAVEATS:
Although overall effects were not found by group over time, additional data analyses will be conducted to determine if there were positive effects for specific subgroups of people.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes